CLINICAL TRIAL: NCT03831087
Title: Cardiac Magnetic Resonance Imaging Versus Computed Tomography to Guide Transcatheter Aortic Valve Replacement: A Randomized Multicenter Trial
Brief Title: Cardiac Magnetic Resonance Imaging Versus Computed Tomography to Guide Transcatheter Aortic Valve Replacement
Acronym: TAVR-CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Johannes Kepler University of Linz (Other); Klinikum Wels-Grieskirchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20171002-1653
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVR-CMR (Other): All MR examinations will be performed with a 1.5-T clinical MR imaging unit (AVANTO_fit; Siemens, Erlangen, Germany). The MR protocol consists of a Navigator-gated free breathing 3D "whole-heart" coronary magnetic resonance angiography (MRA), axial 2D true fast imaging with steady-state free precession (true-FISP) during free breathing covering whole body trunk and a coronal 3D fast low-angle shot (FLASH) Gd-MRA.
  Interventions: Diagnostic Test: TAVR-CMR
- TAVR-CT (Other): All CT examinations will be performed on a 128-slice dual-source CT and high-pitch factor. Prospective electrocardiographic synchronization will be applied, triggered into the diastolic phase for the heart. An injected bolus of 70 to 110 mL of nonionic iodine contrast agent will be applied with 370 mg/mL iodine concentration, using an automatic injector at a flow rate of 5 mL/s, followed by 40 mL saline solution. Contrast agent volume for each patient will be calculated by scan time and body weight. Patients will be placed supine with arms overhead. The scan length range from supraaortic branches to the groins.
  Interventions: Diagnostic Test: TAVR-CT

INTERVENTIONS:
Diagnostic Test: TAVR-CMR — CMR protocol for the exact determination of the aortic valve dimensions, valve size and implantation route.
  Arms: TAVR-CMR
Diagnostic Test: TAVR-CT — CT protocol for the exact determination of the aortic valve dimensions, valve size and implantation route.
  Arms: TAVR-CT

SUMMARY:
To prove the non-inferiority of TAVR-CMR compared to TAVR-CT to guide TAVR according to clinical efficacy, defined as implantation success based on the VARC-2 criteria.

DETAILED DESCRIPTION:
Study Title: Cardiac Magnetic Resonance Imaging Versus Computed Tomography to Guide Transcatheter Aortic Valve Replacement (TAVR-CMR).

Coordinating Prinicpal Investigator: Prof. Bernhard Metzler, University Clinic of Internal Medicine III, Cardiology and Angiology, Innsbruck Medical University.

Planned Study Period: 2017-2023.

Objective: To investigate, for the first time, the non-inferiority of TAVR-CMR to contrast-enhanced computed tomography (TAVR-CT) regarding efficacy and safety end-points.

Design: Prospective, randomized, open-label, multi-centre trial.

Patients (planned): 270 patients.

Diagnosis / Inclusion Criteria: Symptomatic severe aortic stenosis scheduled for TAVR based on a local heart-team decision.

Methods: Patients will be randomized in a 1:1 fashion to receive a predefined TAVR-CMR protocol or to receive a standard TAVR-CT protocol within two weeks after inclusion.

Main Outcome Measure: Follow-up will be performed at hospital discharge after TAVR and after 6 months. The primary efficacy outcome is device implantation success at discharge. The secondary endpoints are a combined safety endpoint and a combined clinical efficacy endpoint at baseline and at 6 months, as well as a comparison of imaging procedure related variables (see section 5.11.2). Endpoint definitions are based on the updated 2012 VARC-2 consensus document.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Severe aortic stenosis according to recent guidelines (aortic valve area ≤ 1.0cm² or aortic valve index ≤ 0.6 cm²/m²) (1)
3. Typical symptoms of severe aortic stenosis like shortness of breath, angina or syncope
4. Patient is evaluated for TAVR

Exclusion Criteria:

1. Contraindications to perform CMR
2. Contraindications to perform CT
3. Contraindications for TAVR or reduced life expectancy < 1 year.
4. Known hypersensitivity to CMR or CT contrast agents
5. Childbearing potential or inability to exclude pregnancy
6. Inability to understand and follow study-related instructions
7. Severe renal insufficiency requiring renal replacement therapy
8. Severe hepatic insufficiency (Child-Pugh class B or C)
9. Post organ transplantation
10. Participation in another clinical study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
The non-inferiority of TAVR-CMR compared to TAVR-CT to guide TAVR according to clinical efficacy, defined as implantation success based on the VARC-2 criteria. | 6 months
  The primary outcome will be a composite clinical efficacy end-point related to implantation success at hospital discharge, based on the VARC-2 criteria: Absence of procedural mortality AND correct positioning of the prosthetic valve AND intended performance of the prosthetic valve (mean aortic valve gradient < 20mmHg and no valve regurgitation > mild)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Metzler, Prof., Principal Investigator — Medical University Innsbruck
Locations (1):
- University Clinic of Internal Medicine III, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lechner I, Oberhollenzer F, Tiller C, Holzknecht M, Kaser A, Binder RK, Gollmann-Tepekoylu C, Klug G, Mayr A, Bauer A, Metzler B, Reindl M, Reinstadler SJ. Age and sex-related outcomes in cardiovascular magnetic resonance versus computed tomography-guided transcatheter aortic valve replacement: a secondary analysis of a randomized clinical trial. J Cardiovasc Magn Reson. 2025 Summer;27(1):101882. doi: 10.1016/j.jocmr.2025.101882. Epub 2025 Mar 13. PMID 40089160
- [Derived] Reindl M, Lechner I, Holzknecht M, Tiller C, Fink P, Oberhollenzer F, von der Emde S, Pamminger M, Troger F, Kremser C, Lassnig E, Danninger K, Binder RK, Ulmer H, Brenner C, Klug G, Bauer A, Metzler B, Mayr A, Reinstadler SJ. Cardiac Magnetic Resonance Imaging Versus Computed Tomography to Guide Transcatheter Aortic Valve Replacement: A Randomized, Open-Label, Noninferiority Trial. Circulation. 2023 Oct 17;148(16):1220-1230. doi: 10.1161/CIRCULATIONAHA.123.066498. Epub 2023 Aug 27. PMID 37634187
- [Derived] Klug G, Reinstadler S, Troger F, Holzknecht M, Reindl M, Tiller C, Lechner I, Fink P, Pamminger M, Kremser C, Ulmer H, Bauer A, Metzler B, Mayr A. Cardiac magnetic resonance imaging versus computed tomography to guide transcatheter aortic valve replacement: study protocol for a randomized trial (TAVR-CMR). Trials. 2022 Sep 2;23(1):726. doi: 10.1186/s13063-022-06638-6. PMID 36056444